CLINICAL TRIAL: NCT05509296
Title: A Prospective, Multicenter, Randomized Control, Non-inferiority to Investigate the Effectiveness and Safety of SINOMED CBC for Endovascular Treatment of Stenotic Coronary Artery Disease
Brief Title: Compare the Effectiveness and Safety of Two Different Kinds of Cutting Balloon in Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sino Medical Sciences Technology Inc. (Industry)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SN-CBC-202201
Record Dates: First submitted 2022-08-16; First posted 2022-08-22 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Coronary Stenosis; Coronary Artery Stenosis; In-stent Restenosis
Keywords: Coronary dilation catheter; Percutaneous coronary artery dilatation; Restenosis; Cutting balloon catheter; scoring balloon catheter
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, randomized control,non-inferiority clinical study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SINOMED CBC (Experimental): Cutting balloon catheter (Sino Medical Sciences Technology Inc.)
  Interventions: Device: SINOMED CBC
- NSE Coronary Dilatation Catheter (Active Comparator): NSE Coronary Dilatation Catheter (Goodman Co.,Ltd)
  Interventions: Device: NSE Coronary Dilatation Catheter

INTERVENTIONS:
Device: SINOMED CBC — The Coronary Dilatation Balloon Catheter is indicated for the treatment of hemodynamically significant coronary artery stenosis, including in-stent restenosis and complex type C lesions, for the purpose of improving myocardial perfusion.
  Other Names: cutting balloon catheter; scoring balloon catheter
  Arms: SINOMED CBC
Device: NSE Coronary Dilatation Catheter — The Coronary Dilatation Balloon Catheter is indicated for the treatment of hemodynamically significant coronary artery stenosis, including in-stent restenosis and complex type C lesions, for the purpose of improving myocardial perfusion.
  Other Names: Lacrosse NSE
  Arms: NSE Coronary Dilatation Catheter

SUMMARY:
The objective of this study is to evaluate safety and effectiveness of the SINOMED CBC coronary dilatation catheter during PCI in subjects with stenotic coronary arteries.

DETAILED DESCRIPTION:
The investigation is a prospective, multi-center, randomized control, non-inferiority clinical study. The study will be conducted in up to 8 investigational sites in the China This study will enroll and treat 136 subjects, including in-stent restenosis (ISR). The population for this study is subjects with stenotic coronary artery disease who are suitable candidates for PTCA.

After screening for initial inclusion and exclusion criteria, eligible subjects will be asked to participate in the study by signing a consent form. Following consent, subjects will undergo a baseline visit where eligibility criteria will be assessed. Then, subjects will be randomized to either trial balloon (Sino Medical Sciences Technology Inc. ) or to a NSE Coronary Dilatation Catheter (Goodman Co.,Ltd). Angiograms will be performed before and after intervention.

Subjects will be followed through hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is at least 18 to 75 years of age, male or not pregnant female.
2. Evidence of myocardial ischemia without symptoms, stable or unstable angina, silent ischemia demonstrated by positive territorial functional study, or old myocardial infarction.
3. De novo or restenotic lesion(s) in native coronary arteries, including in-stent restenosis.
4. Reference vessel diameter (RVD) must be visually estimated ≥ 2.5 and ≤ 5.0mm, and the vessel length must be no more than 30mm.
5. Target lesion(s) must have a diameter stenosis of (a) ≥70% by visual estimation or (b) >50% with evidence of ischemia.
6. The patient has a planned intervention at no more than two de novo lesions, in different epicardial vessels.
7. Investigators believe that target lesion atherosclerotic plaques require spinous balloon treatment and balloon can be passed through by pre-dilation.
8. Able to understand the purpose of the trial, voluntarily participate and sign the informed consent.

Exclusion Criteria:

1. Evidence of ongoing acute myocardial infarction within a week.
2. Chronic total occlusion (TIMI 0), left main lesion, intervention-required three-vessel lesions, and bypass lesion.
3. Severe calcification and Target lesion in a severe angulation (> 45 degrees).
4. Patient has serious heart failure symptoms (NYHA level III or IV), or Left ventricular ejection fraction (LVEF) <40%.
5. Patient with renal dysfunction, as Cr>176.82umol/L or Cr >2.0 mg/dl.
6. Patient with active gastrointestinal bleeding history, any other evidence based bleeding, such as suspected liver failure disease, suffered from cerebral bleeding history, stroke during the last 6 months, with contra-indication of anti-platelet or anti-coagulation.
7. Patients with allergies to heparin and contrast media.
8. Target lesion demonstrating severe dissection prior to planned deployment of the trial device.
9. Visible thrombus at the target lesion.
10. Patients received heart transplantation.
11. Participation in another clinical trial (12 months after index procedure).
12. Those who participated in another clinical trials, but did not reach the primary endpoint.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Rate of Device procedural success (lesion level) | immediate post-intervention(approximately 1.4 hour)
  Defined as: Successful delivery, inflation, deflation, and withdrawal of the study balloon; and ≤30% final diameter stenosis following completion of the interventional procedure, including adjunctive stenting (For ISR or DCB related stenosis, Final diameter stenosis<50%)

SECONDARY OUTCOMES:
Rate of Procedural success (patient level) | during the hospital stay, an average of 7 days post-procedure
  Defined as: ≤30% final diameter stenosis following completion of the interventional procedure, including adjunctive stenting (For ISR or DCB related stenosis, Final diameter stenosis<50%); and freedom from major adverse cardiac events (MACE) during hospitalization
Rate of Target lesion failure (TLF) | during the hospital stay, an average of 7 days post-procedure
  a composite of cardiac death, target vessel myocardial infarction, or clinically-driven target lesion revascularisation (CI-TLR)
Rate of Patient-oriented composite endpoint (POCE) | during the hospital stay, an average of 7 days post-procedure
  a composite of all-cause death, any stroke, any myocardial infarction, or any clinically, and physiologically driven revascularization
Incidence of any AE and SAE incidence | during the hospital stay, an average of 7 days post-procedure
  report any AE results from a device deficiency or other device issue as related to the use of the study device. Such as Balloon burst、vascular perforation, dissection, acute occlusion, vasospasm, thrombosis (including stent thrombosis), arrhythmia requiring intervention, and so on.
Rate of device defect | during the hospital stay, an average of 7 days post-procedure
  report any device defect during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: jianping li, M.D/Ph.D, Principal Investigator — Peking University First Hospital
Locations (8):
- China (8):
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Kaifeng Central Hospital, Kaifeng
  - The First People's Hospital of Lianyungang, Lianyungang
  - Tianjin Chest Hospital, Tianjin
  - Tianjin Forth Central Hospital, Tianjin
  - Wuxi People's Hospital, Wuxi
  - Xuzhou cancer hospital, Xuzhou